CLINICAL TRIAL: NCT00518804
Title: Functional Behavioural Skill Training for Young Children With Severe Autism
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hamilton Health Sciences Corporation (Other)
Responsible Party: Dr. Jo-Ann Reitzel, McMaster University
Organization: McMaster University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Reitzel 2007
Record Dates: First submitted 2007-08-17; First posted 2007-08-21 (Estimated); Last update posted 2008-12-05 (Estimated); Status verified 2008-07

CONDITIONS: Autistic Disorder
MeSH Terms: conditions — Autistic Disorder

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Functional Behavioural Skills Group and Parent Training

SUMMARY:
LAY SUMMARY:

IBI is costly and there are currently long waitlists of children who are in need of treatment. The investigators have clinical and ethical obligations to determine more appropriate alternatives to IBI for children making few gains because all children with autism deserve treatment based on their needs. This study is designed to determine the effectiveness of a functional skills group intervention, based on the principles of applied behaviour analysis, for children responding slowly to IBI. Specifically, it will investigate the effectiveness of functional behavioural skills training in addition to IBI at increasing a child's independence in day to day communication and self-help skills and reducing behaviour problems, as well as increasing parental competence and decreasing caregiver strain compared with IBI alone. Having an effective alternative to IBI for children making few gains is relevant from the standpoint of i) preventing exposure to potentially intrusive interventions for those children making few gains in IBI, ii) allowing children making few gains in IBI to access effective treatment, iii) opening limited IBI spots for children who would benefit from IBI, and iv) making better use of limited health resources. Overall, the results will be of interest to parent, clinicians, researchers and funding bodies.

HYPOTHESES

Four main hypotheses are presented to examine the effectiveness of involvement in the ABA functional skills group in improving parent training and functional skills and behaviour in young children with ASD who do not master the ELM. We focus our hypotheses on child measures of functional self help skills, behaviour and cognition as well as parental measures of caregiver strain and sense of competence.

Participants (i.e. children predicted to have poor response to IBI alone) who attend the functional skills group for 8 months will have:

1. greater decreases in interfering behaviour as measured on the Developmental Behaviour Checklist and ratings of behaviour during observations compared to children receiving IBI alone.
2. greater increases in self-help as measured on the Vineland Adaptive Behaviour Scales II, and greater independence in eating, toileting, requesting, hand washing, and responding to name as measured by independent ratings of these skills compared with those children receiving IBI alone.
3. parents of these children will have greater improvements in their sense of competence as a parent and greater reductions in caregiver strain, compared with parents of children receiving IBI alone.
4. a similar pattern of little or no change in cognitive function compared with children who receive only IBI based on the Stanford Binet. In other words, there will be no difference between the experimental and control group on the measure of cognitive functioning

ELIGIBILITY:
Inclusion Criteria:

* Children receiving Intensive Behavioural Intervention from the Hamilton Niagara Regional Early Autism Intervention Program who do not master the Early Learning Measure after 4 months of treatment

Exclusion Criteria:

* Children receiving Intensive Behavioural Intervention from the Hamilton Niagara Regional Early Autism Intervention Program who master the Early Learning Measure after 4 months of treatment

Ages: 3 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 32 (Estimated)
Dates: Start 2007-08; Study Completion 2009-08 (Estimated)

PRIMARY OUTCOMES:
Parenting Sense of Competence | Before entry to and upon exit from the intervention
Child Behavioural Skills Assessment | Before entry to and upon exit from the intervention

SECONDARY OUTCOMES:
Child Intellectual Functioning | Before entry to and upon exit from the intervention
Child Language Functioning | Before entry to and upon exit from the intervention
Child Adaptive Behaviour | Before entry to and upon exit from the intervention
Child Maladaptive Behaviour | Before entry to and upon exit from the intervention
Caregiver Strain | Before entry to and upon exit from the intervention
Parent Behaviour Skills Assessment | Before entry to and upon exit from the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Jo-Ann Reitzel, PhD., Principal Investigator — McMaster University, Department of Psychiatry and Behavioural Neurosciences
Locations (1):
- McMaster University, 1280 Main Street West, Hamilton, Ontario, Canada